CLINICAL TRIAL: NCT04884035
Title: A Phase 1b, Open Label, Global, Multicenter, Dose Determination, Randomized Dose Expansion Study to Determine the Maximum Tolerated Dose, Assess the Safety and Tolerability, Pharmacokinetics and Preliminary Efficacy of Iberdomide (CC-220) in Combination With R-CHOP-21 and CC-99282 in Combination With R-CHOP-21 for Subjects With Previously Untreated Aggressive B-cell Lymphoma
Brief Title: Study of Safety and Efficacy of Iberdomide (CC-220) and CC-99282 Combined With R-CHOP to Treat Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-DLBCL-001; 2020-005705-71 (EudraCT Number)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma, B-Cell
Keywords: Iberdomide; CC-220; CC-99282; Phase 1; B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — iberdomide; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Administration of CC-220 with R-CHOP-21 (Experimental): CC-220 to be administered orally in combination with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (R-CHOP-21) for 6 cycles of treatment
  Interventions: Drug: CC-220; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Administration of CC-99282 with R-CHOP-21 (Experimental): CC-99282 to be administered orally in combination with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (R-CHOP-21) for 6 cycles of treatment
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: CC-99282
- Administration of CC-220 with polatuzumab-R-CHP (Experimental): CC-220 to be administered orally in combination with Polatuzumab vedotin, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone (polatuzumab-R-CHP) for 6 cycles of treatment
  Interventions: Drug: CC-220; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Polatuzumab vedotin; Drug: Rituximab
- Administration of CC-99282 with polatuzumab-R-CHP (Experimental): CC-99282 to be administered orally in combination with Polatuzumab vedotin, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone (polatuzumab-R-CHP) for 6 cycles of treatment
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: CC-99282; Drug: Polatuzumab vedotin; Drug: Rituximab

INTERVENTIONS:
Drug: CC-220 — CC-220 by mouth at the assigned dose starting on Day 1 for 14 consecutive days of the 21-day treatment cycle for 6 cycles of treatment.
  Other Names: Iberdomide; BMS-986382
  Arms: Administration of CC-220 with R-CHOP-21; Administration of CC-220 with polatuzumab-R-CHP
Drug: Rituximab — Rituximab 375 mg/m2 on Day 1 by intravenous (IV) infusion or 1400 mg (SC) subcutaneous (from Cycle 2) of a 21-day treatment cycle for up to a total of 6 cycles
  Arms: Administration of CC-220 with R-CHOP-21; Administration of CC-99282 with R-CHOP-21
Drug: Cyclophosphamide — Cyclophosphamide 750mg/m2 on Day 1 by IV infusion of a 21-day treatment cycle for up to a total of 6 cycles
Drug: Doxorubicin — Doxorubicin 50 mg/m2 IV infusion on Day 1 of a 21-day treatment cycle for up to a total of 6 cycles
Drug: Vincristine — Vincristine 1.4 mg/m2 (maximum of 2.0 mg total) IV intravenous on Day 1 of a 21-day treatment cycle for up to a total of 6 cycles
  Arms: Administration of CC-220 with R-CHOP-21; Administration of CC-99282 with R-CHOP-21
Drug: Prednisone — Prednisone 100 mg PO on Days 1 through 5 of each 21-day treatment or 100mg IV on Day 1 is also acceptable for up to a total of 6 cycles
  Other Names: Prednisolone
Drug: CC-99282 — CC-99282 by mouth at the assigned dose starting on Day 1 for 7 consecutive days of the 21-day treatment cycle for 6 cycles of treatment.
  Other Names: BMS-986369
  Arms: Administration of CC-99282 with R-CHOP-21; Administration of CC-99282 with polatuzumab-R-CHP
Drug: Polatuzumab vedotin — Polatuzumab vedotin 1.8 mg/kg on Day 1 by intravenous (IV) infusion of a 21-day treatment cycle for up to a total of 6 cycles
  Arms: Administration of CC-220 with polatuzumab-R-CHP; Administration of CC-99282 with polatuzumab-R-CHP
Drug: Rituximab — Rituximab 375 mg/m2 on Day 1 by intravenous (IV) infusion of a 21-day treatment cycle for up to a total of 6 cycles
  Arms: Administration of CC-220 with polatuzumab-R-CHP; Administration of CC-99282 with polatuzumab-R-CHP

SUMMARY:
This is a Phase 1b study consisting of 2 parts: a dose escalation (Part 1) of CC-220 or CC-99282 added to the standard R-CHOP-21 regimen for first-line treatment of a-BCL. The dose escalation (Part 1) will consist of 2 parallel arms in combination with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP-21); CC-220 and R-CHOP-21 or CC-99282 and R-CHOP-21. Part 1 will be followed by a randomized dose expansion (Part 2) with CC-220 and/or CC-99282 at the Recommended Phase 2 Dose (RP2D) in combination with R-CHOP-21. A polatuzumab-R-CHP regimen in combination with CC-220 or CC-99282 will be explored with the addition of a new cohort only after the RP2D for the CC-220 and/or CC-99282 and R-CHOP-21 combination has been defined.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy the following criteria to be enrolled in the study:

  1. Is ≥ 18 years of age at the time of signing the informed consent form (ICF).
  2. Participant has histologically confirmed (per local evaluation) diagnosis of de novo, previously untreated, a-BCL according to 2016 WHO classification.
  3. Participant has International Prognostic Index (IPI) score 0-5 in Part 1 and IPI 2-5 in Part 2. For the CELMoD and polatuzumab-R-CHP cohort, the subject must also have IPI score 0 to 5 in Part 2A and IPI 2 to 5 in Part 2B.
  4. Participants must have measurable disease defined by at least one FDG-avid lesion for FDG-avid subtype and one bi-dimensionally measurable (> 1.5 cm in longest diameter) disease by computed tomography (CT) or magnetic resonance imaging (MRI), as defined by the Lugano classification (Cheson, 2014).
  5. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
  6. Participants must have the following laboratory values:

     1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L or ≥ 1.0 x 109/L in case of documented bone marrow involvement (> 50% or tumor cells), without growth factor support for 7 days (14 days if peg-G-CSF)
     2. Hemoglobin (Hb) ≥ 8 g/dL
     3. Platelets (PLT) ≥ 75 x 109/L or ≥ 50 x 109/L in case of documented bone marrow involvement (>50% or tumor cells), without transfusion for 7 days
     4. Aspartate aminotransferase / serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase / serum glutamate pyruvic transaminase (ALT/SGPT) ≤ 2.5 x upper limit of normal (ULN). In the case of documented liver involvement by lymphoma, ALT/SGPT and AST/SGOT must be ≤ 5.0 x ULN.
     5. Serum total bilirubin ≤ 2.0 mg/dL except in cases of Gilbert's syndrome, then ≤ 5.0 mg/dl. Subjects receiving polatuzumab vedotin must have serum total bilirubin < 1.5 × ULN (26 μmol/L) (corresponding to mild degree as per National Cancer Institute Organ Dysfunction Working Group [NCI ODWG] criteria) except in cases of Gilbert's syndrome, then ≤ 3.0 mg/dl (51 μmol/L).
     6. Estimated serum creatinine clearance (CrCl) of ≥ 50 mL/min using the modification of diet in renal disease (MDRD) formula.
  7. All participants must:

     1. Have an understanding that the study drug could have a potential teratogenic risk.
     2. Agree to follow all requirements defined in the Pregnancy Prevention Program for CC-220 or CC-99282 Pregnancy Prevention Plan for Participants in Clinical trials.
  8. Females of childbearing potential (FCBP) must:

     a. Have two negative pregnancy tests as verified by the investigator prior to starting study therapy.
  9. Male participants must:

     1. Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study.

Exclusion Criteria:

* The presence of any of the following will exclude a participant from enrollment:

  1. Any significant medical condition, active infection (including SARS-CoV-2 suspected or confirmed), laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
  2. Any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
  3. Any other subtype of lymphoma.
  4. Documented or suspected CNS involvement by lymphoma.
  5. Persistent diarrhea or malabsorption ≥ Grade 2 (NCI CTCAE v5.0), despite medical management.
  6. Peripheral neuropathy ≥ Grade 2 (NCI CTCAE v5.0).
  7. Subjects with a history of progressive multifocal leukoencephalopathy.
  8. Chronic systemic immunosuppressive therapy or corticosteroids
  9. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

     a. Left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO)
  10. Major surgery ≤ 2 weeks prior to starting CC-220 or CC-99282; participant must have recovered from any clinically significant effects of recent surgery.
  11. Any condition causing inability to swallow tablets.
  12. Known seropositivity for or active viral infection with human immunodeficiency virus (HIV)
  13. Known chronic active hepatitis B (hepatitis B virus surface antigen [HBsAg] positive and/or hepatitis B core antibody [anti-HBc] positive with viral DNA positive) or C (positive serology requiring treatment and/or with evidence of liver damage) infection
  14. History of other malignancy, unless being free of the disease for ≥ 3 years; exceptions to the ≥ 3-year time limit include history of the following:

      1. Localized nonmelanoma skin cancer
      2. Carcinoma in situ of the cervix
      3. Carcinoma in situ of the breast
      4. Incidental histologic finding of prostate cancer (T1a or T1b as per Tumor Node Metastasis [TNM] staging system) or prostate cancer that has been treated with curative intent.
  15. Hypersensitivity to the active substance or to murine proteins, or to any of the other excipients of rituximab or polatuzumab vedotin.
  16. Known hypersensitivity to any component of CHOP/CHP regimen.
  17. Known allergy to thalidomide, pomalidomide, or lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) - Part 1 | During the first 2 cycles of treatment (each cycle is 21 days)
  Frequency of dose-limiting toxicities (DLT) associated with addition of iberdomide (CC-220) to R-CHOP-21 therapy and the addition of CC-99282 to R-CHOP-21 therapy
Recommended Phase 2 Dose (RP2D) - Part 1 | During the first cycle of treatment (each cycle is 21 days)
  Defined as the dose that will be selected for dose expansion based on MTD
Safety and tolerability of CC-220 and CC-99282 at RP2D - Part 2 | From the first dose of any IP until 28 days after the last dose of IP
  AEs evaluated using NCI CTCAE criteria, v. 5.0, including treatment -emergent adverse events (TEAEs) and laboratory assessments
Maximum Tolerated Dose (MTD) - Part 2A | During the first cycle of treatment (each cycle is 21 days)
  Frequency of DLTs associated with addition of iberdomide (CC-220) to polatuzumab-R-CHP therapy and the addition of CC-99282 to polatuzumab-R-CHP therapy
Recommended Phase 2 Dose (RP2D) - Part 2A | During the first cycle of treatment (each cycle is 21 days)
  Defined as the dose that will be selected for dose expansion based on MTD

SECONDARY OUTCOMES:
Best overall response rate (ORR) | Up to 4 years
  The proportion of participants with best overall response achieved during the study as either Complete Response or Partial Response before subsequent anti-lymphoma therapy
Complete Metabolic Response Rate (CMRR) | Up to 4 years
  The proportion of participants experiencing complete metabolic response (CMR) before receiving any subsequent anti-lymphoma therapy
Time to Response (TTR) | Up to 4 years
  The time from entry to the study (enrollment date for Part 1 and randomization date for Part 2) to the date of first documented response (≥ PR)
Duration of Response (DOR) | Up to 4 years
  The time from the earliest date of documented response (≥ PR) to the first occurrence of relapse or progression
Progression-free Survival (PFS) | Up to 4 years
  The time from entry to the study (enrollment date for Part 1 and randomization date for Part 2) to the first occurrence of disease progression or death from any cause
Overall Survival (OS) | Up to 4 years
  The time from entry to the study (enrollment date for Part 1 and randomization date for Part 2) to death from any cause
Pharmacokinetics - Cmax for CC-220 | At Cycle 1 Day 7, Cycle 1 Day 15, and Cycle 2 Day 7 (each cycle is 21 days)
  Maximum plasma concentration of drug
Pharmacokinetics - Ctrough for CC-220 | At Cycle 1 Day 7, Cycle 1 Day 15, and Cycle 2 Day 7 (each cycle is 21 days
  Minimum or trough concentration
Pharmacokinetics - Tmax for CC-220 | At Cycle 1 Day 7, Cycle 1 Day 15, and Cycle 2 Day 7 (each cycle is 21 days
  Time to maximum plasma concentration
Pharmacokinetics - Cmax for CC-99282 | At Cycle 1 Day 7, Cycle 1 Day 15, and Cycle 2 Day 7 (each cycle is 21 days
  Maximum plasma concentration
Pharmacokinetics - Ctrough for CC-99282 | At Cycle 1 Day 7, Cycle 1 Day 15, and Cycle 2 Day 7 (each cycle is 21 days
  Minimum or trough concentration
Pharmacokinetics - Tmax for CC-99282 | At Cycle 1 Day 7, Cycle 1 Day 15, and Cycle 2 Day 7 (each cycle is 21 days
  Time to maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (40):
- United States (14):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Local Institution - 169, Duarte, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center Of Kansas-Wichita, Wichita, Kansas
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - HealthPartners Cancer Research Center, Saint Louis Park, Minnesota
  - University of Nebraska - Fred and Pamela Buffet Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Local Institution - 170, Charlotte, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 168, Murray, Utah
  - Local Institution - 171, St. George, Utah
- Australia (3):
  - Local Institution - 501, Adelaide, South Australia
  - Local Institution - 503, Perth
  - Local Institution - 502, Waratah
- Greece (5):
  - Evangelismos General Hospital of Athens, Athens
  - General Hospital of Athens "Laiko", Athens
  - Attikon University General Hospital, Athens
  - Local Institution - 703, Pátrai
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Poland (8):
  - AIDPORT Sp. z o.o., Skórzewo, Greater Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - MCM Krakow - PRATIA - PPDS, Krakow
  - Local Institution - 0706, Poznan
  - Local Institution - UNK0706, Poznan
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Słomniki
  - Local Institution - 602, Warsaw
  - Local Institution - 604, Wroclaw
- South Korea (3):
  - Local Institution - 300, Seoul
  - Local Institution - 302, Seoul
  - Local Institution - 301, Seoul
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol ICO Badalona, Barcelona
  - Local Institution - 204, Madrid
  - H. Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04884035.html